CLINICAL TRIAL: NCT03517189
Title: Hemodynamic Changes During Displacement of the Heart in the Aorta No-touch Off-pump Coronary Artery Bypass Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Solange Guizilini, Principal Investigator, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63054016.1.0000.5505
Record Dates: First submitted 2018-04-12; First posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Cardiac Surgery; Aorta No-touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aorta no-touch (Experimental): Aorta no-touch off-pump coronary artery bypass surgery.
  Interventions: Procedure: Aorta no-touch

INTERVENTIONS:
Procedure: Aorta no-touch — Participants will be submitted to aorta no-touch off-pump coronary artery bypass surgery.

SUMMARY:
Introduction: Aorta no-touch off-pump coronary artery bypass surgery (OPCAB) has been the recommended technique for treatment of patients with high-risk of neurological damage or stroke. However, the displacement of the heart to achieve suitable exposure for graft construction elicits hemodynamic changes, potentially requiring conversion to on-pump. Objective: The aim of this study is to evaluate the sequential changes of hemodynamic parameters in patients that undergo aorta no-touch OPCAB. Method: Patients that undergo aorta no-touch OPCAB will be evaluated. The FloTrac / PreSep / Vigileo ™ (Edwards Lifesciences) system will be used to continuously record heart rate (HR), mean arterial pressure (DBP), central venous pressure (CVP), continuous cardiac index, systolic volume , systolic volume variation (VVS) and central venous oxygen saturation (ScvO2). The parameters will be evaluated 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending PD, marginal-OM and diagonal-Dg). Postoperative lactate will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of coronary artery disease with indication of myocardial revascularization surgery

Exclusion Criteria:

* patients will be excluded if they presented clinically significant preoperative hepatic or renal dysfunction, thrombocytopenia, coagulopathy, or uncontrolled arrhythmia.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in heart rate | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac/PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in heart rate during procedures
Change in mean arterial blood pressure | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac/PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in mean arterial blood pressure during procedures
Change in central venous pressure | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac/PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in central venous pressure during procedures
Change in continuous cardiac index | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac/PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in continuouns cardiac index during procedures
Change in stroke volume | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac/PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in stroke volume during procedures
Change in central venous oxygen saturation | The parameters will be assessed 5 min before, during and 5 min after each anastomosis (left anterior descending-LAD, posterior descending-PD, marginal-OM and diagonal-Dg).
  By the FloTrac /PreSep/Vigileo™ system (Edwards Lifesciences), assessing the change in central venous oxygen saturation during procedures

SECONDARY OUTCOMES:
Evaluate lactate levels | Immediate postoperative period, at the admission on the intensive care unit
  Evaluation of the lactate levels in the immediate postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No